CLINICAL TRIAL: NCT00897429
Title: Correlative Science Studies in Colon Cancer a Companion Study to CALGB 9581 and 89803
Brief Title: Studying Tissue Samples From Patients With Stage II Colon Cancer Treated on Clinical Trial CLB-9581
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-150705; CDR0000559812 (Registry Identifier: NCI Physician Data Query); NCI-2009-00452 (Registry Identifier: NCI Clinical Trial Reporting Program); U10CA180821 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer
Keywords: stage IIA colon cancer; stage IIB colon cancer; stage IIC colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (laboratory biomarker analysis): Previously collected tissue samples are analyzed for K-ras mutations; COX-2, phospho-AKT, and VEGF overexpression; microvessel density; association of genomic instability with microsatellite instability and p53 mutations; and methylation status of MLH1, MGMT, and WRN and to identify prognostic biomarkers by LINE-1 hypomethylation, PIK3CA mutation, BRAF mutation, FASN expression, and VDR expression via immunohistochemistry, PCR, RT-PCR, and microarray.
  Interventions: Procedure: laboratory biomarker analysis

INTERVENTIONS:
Procedure: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies tissue samples from patients with stage II colon cancer treated on Cancer and Leukemia Group B (CALGB)-9581 or CALGB-90903. Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer. It may also help doctors understand how patients respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the impact of loss of p21 and mutations in p53 on the relationship between higher intake of a Western dietary pattern (manifested by higher red meat and total fat intake and lower n-3 polyunsaturated fatty acids, fruit and vegetable intake) and colon cancer recurrence/mortality. (B1)

II. To evaluate the impact of mutated v-Ki-ras2 Kirsten rat sarcoma viral oncogene homolog (K-ras), mutated p53, phorphorylated (phospho)-v-akt murine thymoma viral oncogene homolog 1 (Akt) overexpression, and p27 loss on the relationship between each of obesity, physical activity and dietary glycemic intake and colon cancer recurrence/mortality. (B1)

III. To evaluate the impact of tumoral cyclooxygenase-2 (COX-2) and vascular endothelial growth factor (VEGF) overexpression, high tumor microvessel density and intact p21 on the relationship between aspirin use and colon cancer recurrence. (B1)

IV. To define the association of type and extent of genomic instability with clinical outcome in stage III colon cancers treated with resection and adjuvant chemotherapy (CALGB 89803). (B2)

V. To assess the ability of a prognostic gene expression signature to stratify stage II colorectal cancer patients into those who will experience relapse within five years post surgery (high risk) and those who will experience five-year disease free survival (low risk), without additional treatment. (B3)

VI. To determine whether there is a significant relationship between the risk of recurrence and the continuous 12-gene recurrence score (RS) as measured by the growth hormone insufficiency (GHI) assay of gene expression, using the pre-specified genes and Recurrence Score algorithm. (B4) VII. To determine whether there is a significant relationship between the risk of recurrence and the continuous 15-gene RS2 as measured by the GHI assay of gene expression, using the pre-specified genes and second-generation Recurrence Score algorithm. (B4)

VIII. To assess the methylation status of mutL homolog 1 (MLH1), o-6-methylguanine-DNA methyltransferase (MGMT), and Werner syndrome (WRN) in tumors obtained from patients enrolled in both treatment arms of CALGB 89803. (B5)

IX. Determine the expression of DNA repair pathway proteins assessed by methylation-specific polymerase chain reaction (MSP) assays as well as the expression of DNA repair proteins that are known to interact with these epigenetically silenced DNA repair proteins using validated immunostaining assays. (B5)

X. Recognition of cytosine phosphate guanine (CpG) island methylator phenotype (CIMP) genes. (B5)

XI. To understand the relationship between tumor gene methylation status and epigenetic silencing of DNA repair pathway genes. (B5)

XII. To examine newly identified prognostic biomarkers (long interspersed nucleotide element 1 [LINE-1] methylation, phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha [PIK3CA] mutation, v-raf murine sarcoma viral oncogene homolog B1 [BRAF] mutation, fatty acid synthase [FASN] expression and vitamin D receptor [VDR] expression) in stage III colon cancers (CALGB 89803) with detailed lifestyle, treatment and follow-up data and correlate them with survival. (B6)

SECONDARY OBJECTIVES:

I. To define the association of type and extent of genomic instability with microsatellite instability and p53 mutations, which have previously been characterized in these tumors by Drs. Warren and Bertagnolli. (B2)

II. Associations with other markers will be determined at some future time once they have been characterized by collaborators. (B2)

III. To determine whether the 12-gene RS provides significant information beyond clinical and pathologic measures, including T stage, mismatch repair system (MMR) status, number of lymph nodes examined, tumor grade, and lymphovascular invasion. (B4)

IV. To determine whether the 15-gene RS2 provides significant information beyond the clinical and pathologic measures, including T stage, MMR status, number of lymph nodes examined, tumor grade, and lymphovascular invasion. (B4)

V. To compare the risk of recurrence between the high and low recurrence risk groups based on pre-specified percentile cut-points for the 12-gene RS. (B4)

VI. To compare the risk of recurrence between the high and low recurrence risk groups based on pre-specified percentile cut-points for the 15-gene RS2. (B4)

VII. To determine, for each of a panel of selected new genes (up to 768 genes), whether there is a significant relationship between gene expression and recurrence-free interval (RFI). (B4)

VIII. To define the association of CIMP and methylated genes with other genetic alterations and tumor-specific characteristics. (B5)

IX. To study the influence of diet and other lifestyle factors on cancer recurrence and treatment-related toxicity in patients participating in this trial. (B6)

OUTLINE:

Previously collected tissue samples are analyzed for K-ras mutations; COX-2, phospho-AKT, and VEGF overexpression; microvessel density; association of genomic instability with microsatellite instability and p53 mutations; and methylation status of MLH1, MGMT, and WRN and to identify prognostic biomarkers by LINE-1 hypomethylation, PIK3CA mutation, BRAF mutation, FASN expression, and VDR expression via immunohistochemistry, polymerase chain reaction (PCR), RT-PCR, and microarray.

ELIGIBILITY:
Inclusion Criteria:

* Registration to CALGB 9581 or 89803
* Samples present within the CALGB Pathology Coordinating Office (PCO) or at the institutions providing treatment that are sufficient to meet study aims
* Institutional Review Board (IRB) review and approval at the institution where the laboratory work will be performed is required
* CALGB does not require that a separate consent form be signed for this study:

  * The subject population to be studied in this protocol includes patients selected from either of the following CALGB treatment protocols: CALGB 9581 or 89803; all such patients have signed (or will sign) a written informed consent document meeting all federal, state, and institutional guidelines as part of entry into those trials
  * All samples to be studied are obtained and stored as part of the patient's respective treatment trial; the material and data obtained from the patient's protocol record will be used to obtain appropriate clinical information; in no instance will the patient be contacted directly
  * There should be no physical, psychological, social, or legal risks associated with this study; no invasive procedures are recommended or requested
  * All appropriate and necessary procedures will be utilized to maintain confidentiality; all patients who have had samples submitted for analysis will have their CALGB study number used to identify specimens
  * This study does not require direct patient contact and no specific risk or benefits to individuals involved in the trial are anticipated; it is likely, however, that the information gained will substantially help similar patients in the future

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer registered to CALGB 9581 or 89803
Sampling Method: Non-Probability Sample
Enrollment: 2059 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Analyses of molecular models among patients who completed the diet and lifestyle questionnaire and who provided tumor blocks for analyses (B1) | Up to 5 years
  Using stratified analyses, effect modification by molecular alterations will be assessed. To maintain statistical power, body mass index and physical activity will be categorized into tertiles for the analyses of interactions with tumor molecular alterations. To assess whether the relative effect of an exposure differs according to the presence of the molecular alteration, tests for statistical interaction will be performed by entering into the model the cross-product term of the molecular alteration (as an indicator variable) and the other risk factor for cancer recurrence.
Proportion of patients who are cancer recurrence-free and alive at 4 years, approximating 4-year disease-free survival for the cohort to be 65% (B1) | 4 years
Influence of energy balance on tumor with specific molecular features (B1) | Up to 5 years
Influence of medications on tumors with specific molecular features (B1) | Up to 5 years
Detection of clones associated with overall survival (OS) (B2) | Up to 5 years
  Proper adjustment for multiplicity must be applied.
Recurrence-free interval (RFI) (B3) | up to 5 years
  Will use the Kaplan Meier product-limit estimator.
Clinical validation of the GHI 12-gene recurrence score (B4) | Up to 5 years
  Weighted Cox proportional hazards regression models will be fit and Wald-type test statistics for the model parameters will be constructed using weighted partial likelihood estimates and robust variance estimates.
Clinical validation of the 15-gene second-generation recurrence score (B4) | Up to 5 years
  Weighted Cox proportional hazards regression models will be fit and Wald-type test statistics for the model parameters will be constructed using weighted partial likelihood estimates and robust variance estimates.
Determination of whether the methylated and silenced DNA repair genes, MLH1, WRN, or MGMT, or CIMP colorectal cancers are associated with OS (B5) | Up to 5 years
Expression of newly identified prognostic biomarkers (LINE-1, PIK3CA, BRAF, FASN and VDR) on OS (B6) | Up to 5 years
  Interaction hazard ratios and the Cox model will be used.
Cancer-specific mortality (B6) | Up to 5 years

SECONDARY OUTCOMES:
Detection of clones associated with disease-free survival (DFS) (B2) | Up to 5 years
  Proper adjustment for multiplicity must be applied.
Determination of whether the methylated and silenced DNA repair genes, MLH1, WRN, or MGMT, or CIMP colorectal cancers are associated with DFS (B5)studies | Up to 5 years
MRE11 status of MSI tumors genetic alterations and tumor-specific characteristics | Up to 5 years
  It is also planned to establish whether this correlates with response to the camptothecin-related compound irinotecan hydrochloride.
Evaluation of up to 768 new genes for their relationship with colon cancer recurrence (B4 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Monica Bertagnolli, MD, Study Chair — Brigham and Women's Cancer Center
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States